CLINICAL TRIAL: NCT06566430
Title: PrEP My Way: a Hybrid Type 1 Clinical Effectiveness-implementation Trial to Promote PrEP Persistence Among Young Kenyan Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Kenya Medical Research Institute (Other); Jomo Kenyatta University of Agriculture and Technology (Other); Kenya National AIDS & STI Control Programme (Other); Emory University (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Professor of Medicine, Director of Research, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024P002284
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: HIV/AIDS
Keywords: prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PrEP My Way intervention (Experimental): PrEP My Way is an intervention that involves peer-delivery of a kit containing PrEP and other sexual health services. Participants will be offered PrEP (if HIV-negative) per a point-of-care test, pregnancy testing, vaginal swabs for gonorrhea and chlamydia testing, condoms, and/or self-injection medroxyprogesterone, as desired.
  Prior to randomization, participants will decide which form of PrEP they would like to take (oral FTC/TDF, dapivirine ring, injectable cabotegravir) and adherence support.
  Interventions: Behavioral: PrEP My Way intervention
- PrEP My Way intervention without STI testing (Experimental): PrEP My Way is an intervention that involves peer-delivery of a kit containing PrEP and other sexual health services. Participants will be offered PrEP (if HIV-negative) per a point-of-care test, pregnancy testing, condoms, and/or self-injection medroxyprogesterone, as desired.
  Prior to randomization, participants will decide which form of PrEP they would like to take (oral FTC/TDF, dapivirine ring, injectable cabotegravir) and adherence support.
  Interventions: Behavioral: PrEP My Way intervention without STI testing
- Enhanced standard of care (Experimental): Prior to randomization, participants will decide which form of PrEP they would like to take (oral FTC/TDF, dapivirine ring, injectable cabotegravir).
  Interventions: Behavioral: Enhanced standard of care

INTERVENTIONS:
Behavioral: PrEP My Way intervention — Intervention components may be modified pending the input from Aim 1. As currently planned, the peer delivering the PrEP My Way kit will be trained to provide basic education and support use of the kit components. The peer will also have a smart phone to show an instructional video. Participants will communicate with peers via mobile phones (e.g., SMS, WhatsApp) to arrange for kit delivery at Months 1, 3, 6, 9, and 12 for those choosing the oral or ring formulations of PrEP. If the participant chooses to use injections, she will communicate with the peers to arrange for kit delivery at Months 1, 3, 5, 7, 9, 11, and 12. All deliveries will be made via unmarked vehicles at home or a preferred safe site during reasonable hours. Two-way mobile phone communication will also be used to convey test results and provide on-going support and empowerment. Follow-up with the clinic will occur at Month 12 and as needed (e.g., treatment for positive tests).
  Arms: PrEP My Way intervention
Behavioral: PrEP My Way intervention without STI testing — Intervention components may be modified pending the input from Aim 1. As currently planned, the peer delivering the PrEP My Way kit will be trained to provide basic education and support use of the kit components. This kit will not contain STI testing. The peer will also have a smart phone to show an instructional video. Participants will communicate with peers via mobile phones (e.g., SMS, WhatsApp) to arrange for kit delivery at Months 1, 3, 6, 9, and 12 for those choosing the oral or ring formulations of PrEP. If the participant chooses to use injections, she will communicate with the peers to arrange for kit delivery at Months 1, 3, 5, 7, 9, 11, and 12. All deliveries will be made via unmarked vehicles at home or a preferred safe site during reasonable hours. Two-way mobile phone communication will also be used to convey test results and provide on-going support and empowerment. Follow-up with the clinic will occur at Month 12 and as needed (e.g., treatment for positive tests).
  Arms: PrEP My Way intervention without STI testing
Behavioral: Enhanced standard of care — These participants will receive PrEP (choice of oral, ring, or injection formulation), STI testing, and family planning at the clinic, as requested.
  Arms: Enhanced standard of care

SUMMARY:
PrEP My Way is a novel PrEP delivery system consisting of clinic-based PrEP initiation, followed by peer-delivered kits for HIV self-testing, PrEP refills, vaginal swabs for gonorrhea and chlamydia self-sampling, pregnancy tests, and contraception refills, if desired. Based on Social Cognitive Theory, the overall hypothesis is that PrEP My Way will overcome critical stigma and structural barriers that currently limit PrEP use and thus empower young women to promote their sexual health.

Preliminary testing of PrEP My Way in Kisumu, Kenya found it to be highly feasible and acceptable, but PrEP use as an oral medication was lower than expected. Now that newer PrEP formulations are becoming available, the team is adding choice of PrEP formulation (i.e., oral tenofovir/emtricitabine, injectable cabotegravir-long acting [CAB-LA], or dapivirine ring) as well as choice of adherence support from peers (e.g., SMS [short message service], routine check-ins and/or WhatsApp groups) to the intervention. The study team will then test the effectiveness of the augmented PrEP My Way intervention (with and without testing for gonorrhea and chlamydia due to cost concerns) on PrEP persistence in women with ongoing HIV prevention needs (i.e., self-reported desire for PrEP, self-reported HIV risk, condomless sex, and/or multiple sexual partners). The team will also track implementation, service, and client metrics per Proctor's framework and determine cost-effectiveness of the intervention

DETAILED DESCRIPTION:
1. Augment PrEP My Way to include choice of PrEP formulation (CAB-LA, dapivirine ring, or oral FTC/ TDF) and adherence support. With a Kenyan design firm, the study team will conduct 28 individual interviews and 2 workshops with young women, young men (as sexual partners), caregivers, nurses, and community health workers to adapt the kit, product guides, and delivery systems. The study team will use a nurse-delivered model for injections per Kenya regulations and a peer-delivered model for rings/oral PrEP. The Kenya National AIDS/STI Control Program will review the design to optimize potential uptake and sustainability in routine care.
2. Conduct a type 1 effectiveness-implementation trial of PrEP My Way. The study team will enroll 432 women (age 16-24) in Kisumu, Kenya, and randomize them 1:1:1 to the full intervention vs the intervention without STI testing (i.e., to assess marginal impact of the most costly kit component beyond PrEP) vs enhanced standard of care. Women in the intervention will choose bimonthly (CAB-LA) or quarterly (ring/oral) delivery. The primary outcome will be PrEP persistence by recorded injection (CAB-LA) or drug levels (ring/oral) at 9 months in women with ongoing HIV prevention needs (i.e., self-reported desire for PrEP, self-reported HIV risk, condomless sex, and/or multiple sexual partners). Secondary/additional outcomes will be persistence and adherence at other time points and with alternative definitions of HIV prevention needs, STI (sexually transmitted infection) testing, and family planning use. Investigators will also track implementation, service, and client metrics per Proctor's framework.
3. Determine cost and cost-effectiveness of PrEP My Way. Analysts will conduct micro-costing analyses through time and motion studies and use published cost data, internal reports, and supply-chain data to determine the cost of delivering each PrEP formulation and support option and the marginal cost of STI testing. The team will also estimate the incremental cost-effectiveness ratio in terms of cost per woman with PrEP persistence.

ELIGIBILITY:
Inclusion Criteria:

* young women (age 16-24 years)
* initiating PrEP at the recruitment site (this criterion subsumes all necessary safety assessments for starting PrEP, including HIV-negative status and for those taking FTC/TDF normal renal function and lack of Hepatitis B infection)
* resident in Kisumu County
* phone ownership
* ability to understand KiSwahili, DhoLuo, and/or English

Exclusion Criteria:

* inability to provide informed consent (e.g., intoxication)

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Months of PrEP persistence | 9 months
  We will consider receipt of CAB-LA injections as count data, we will analyze the amount of dapivirine loaded in the ring minus the residual ring level, and we will analyze the TFV-DP concentrations from dried blood spots in those participants who took oral PrEP. Each measure reflects ~8 weeks of drug coverage, such that an equivalent measure is available for all formulations.

SECONDARY OUTCOMES:
Months of prevention-effective persistence | 9 months
  We will consider receipt of CAB-LA injections as count data, we will analyze the amount of dapivirine loaded in the ring minus the residual ring level, and we will analyze the TFV-DP concentrations from dried blood spots in those participants who took oral PrEP. Each measure reflects ~8 weeks of drug coverage, such that an equivalent measure is available for all formulations. Data will only be considered for those reporting ongoing HIV prevention needs.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, MS, Principal Investigator — Director of Research, Center for Global Health
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya